CLINICAL TRIAL: NCT02492763
Title: A Phase IIa, Multicenter, Placebo- and Active-controlled, Randomized, Double-Blind, Clinical Trial to Evaluate the Safety and Efficacy of MK-8521 Compared to Placebo in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Preliminary Study of the Efficacy and Safety of MK-8521 for Type 2 Diabetes (MK-8521-004)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8521-004; MK-8521-004 (Other: Merck protocol number)
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MK-8521 300 μg (Experimental): Participants receive double-blind MK-8521 300 μg daily (QD), subcutaneously, over 12 weeks.
  Interventions: Drug: MK-8521; Drug: Placebo; Drug: Metformin
- MK-8521 180 μg (Experimental): Participants receive double-blind MK-8521 180 μg QD, subcutaneously, over 12 weeks.
  Interventions: Drug: MK-8521; Drug: Placebo; Drug: Metformin
- Placebo (Placebo Comparator): Participants receive matching double-blind placebo, QD over 12 weeks.
  Interventions: Drug: Placebo; Drug: Metformin
- Liraglutide 1.8 mg (Active Comparator): Participants receive open-label 1.8 mg of liraglutide, QD, subcutaneously, over 12 weeks.
  Interventions: Drug: Liraglutide; Drug: Metformin

INTERVENTIONS:
Drug: MK-8521 — Dose strengths: 180 μg QD administered subcutaneously. A 2-step dose escalation regimen [60 μg, 120 μg] over the first 2 weeks is used to achieve the final dose up to 180 μg.); 300 μg QD administered subcutaneously (A 3-step dose escalation regimen [60 μg, 120 μg, 180 μg] over the first 3 weeks is used to achieve the final dose up to 300 μg.
  Arms: MK-8521 180 μg; MK-8521 300 μg
Drug: Placebo — Double dummy matching placebo for the MK-8521 and placebo arms: matching placebo for MK-8521 300 μg QD administered subcutaneously; matching placebo for MK-8521 180 μg QD administered subcutaneously. A dose escalation regimen consistent with that of the MK-8521 300 μg and 180 μg arms of the study; mock escalation will be performed over the first 2 to 3 weeks.
  Arms: MK-8521 180 μg; MK-8521 300 μg; Placebo
Drug: Liraglutide — Dose strength: 1.8 mg QD administered subcutaneously. A 2-step dose escalation regimen (0.6 mg, 1.2 mg) over the first 2 weeks is used to achieve the final dose up to 1.8 mg.
  Other Names: Victoza®
  Arms: Liraglutide 1.8 mg
Drug: Metformin — Metformin immediate release (IR) or metformin extended release (XR) administered ≥1000 mg QD as background therapy

SUMMARY:
This is a multicenter randomized, double-blind, placebo- and active-controlled (liraglutide; Victoza®), parallel-group, clinical trial of MK-8521 in participants with type 2 diabetes mellitus (T2DM) with inadequate glycemic control while on a stable dose of metformin (≥1000 mg/day).

The trial will include a 1-week screening period; at least an 8-week antihyperglycemic agent (AHA) washout period, if required; a 14-week blinded therapy period (which includes single-blind run-in and double-blind therapy); and a 14-day post-treatment visit, 2 weeks after the last dose of investigational product.

The primary hypothesis of the trial is that MK-8521 provides greater reduction in hemoglobin A1C relative to placebo after 12 weeks of once-daily administration in participants with T2DM with inadequate glycemic control on metformin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Have T2DM in accordance with American Diabetes Association guidelines
* Be on metformin monotherapy (>-1000 mg/day: metformin IR or metformin XR) for at least 12 weeks prior to study start with a hemoglobin A1C (A1C) >-7.5 and <-10.5% OR Be on dual therapy with metformin (>-1000 mg/day: dose stable for at least 4 weeks prior to study start) with an A1C of >-7.0% and <-10.0% and a second AHA and be willing to washout the second AHA. Allowable AHAs are dipeptidyl peptidase 4 (DPP-4 inhibitors), alpha-glucosidase inhibitors, sulfonylureas, and glinides.
* Have a body mass index (BMI) ≥23 kg/m^2 and ≤40 kg/m^2
* Is a female who is not of reproductive potential, or is a female of reproductive potential who agrees to avoid becoming pregnant: while receiving study drug and for 14 days after the last dose of study drug

Exclusion Criteria:

* Have a history of type 1 diabetes or a history of diabetic ketoacidosis
* Has a history of other specific types of diabetes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant)
* Has been treated with any gut-derived incretin hormone glucagon-like peptide 1 (GLP-1) receptor agonist (e.g. Byetta™, Victoza™ or investigational agents) within the last 6 months or has had GLP-1 receptor agonist discontinued due to gastrointestinal intolerance or lack of efficacy. Note: treatment with a GLP-1 receptor agonist that was discontinued >6 months prior to study start is not an exclusion if the GLP-1 receptor agonist was discontinued for reasons other than gastrointestinal intolerance or lack of efficacy.
* Has a history of clinically significant gastrointestinal disorder (including diabetic gastroparesis; irritable bowel disease; recurrent episodes of nausea, vomiting, diarrhea and abdominal pain)
* Has a history of clinically significant and active, immunological, respiratory, genitourinary or major neurological (including stroke, transient ischemic attack and chronic seizures) abnormalities or diseases
* Has a history of cardiovascular disease (including diabetic cardiomyopathy) or significant cardiac condition (including a history of myocardial infarction, stable or unstable angina, arterial revascularization, pathologic, symptomatic or sustained tachyarrhythmia [e.g. atrial fibrillation, sustained supraventricular tachycardia, symptomatic non-sustained supraventricular tachycardia, ventricular tachycardia, ventricular fibrillation, Wolf-Parkinson-White syndrome, congenital long QT syndrome, etc.]) or heart failure
* Has a family history of medullary carcinoma of the thyroid or multiple endocrine neoplasm type-2 syndrome
* Has active diabetic proliferative retinopathy or a history of maculopathy
* Has human immunodeficiency virus (HIV)
* Has a medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic hepatitis B or C (assessed by medical history), primary biliary cirrhosis, or active symptomatic gallbladder disease
* Is on a weight loss medication or has undergone bariatric surgery
* Has a history of acute or chronic pancreatitis of any etiology
* Had an event of severe hypoglycemia with neuroglycopenia in the past 12 months
* Has a positive urine pregnancy test
* Is pregnant or breast-feeding, or is planning to conceive during the trial, including 14 days following the last dose of investigational product
* Routinely consumes >1 alcoholic drinks per day or >7 alcoholic drinks per week or engages in binge drinking
* Routinely consumes ≥480mg /day caffeine in caffeinated beverages (1 cup of coffee contains approximately 120 mg of caffeine
* Is taking a beta blocker or medications with sympathomimetic activity (e.g. pseudoephedrine, phenylpropanolamine, etc.)
* Is currently a user of nicotine or nicotine containing products or does not agree to refrain from using nicotine during the trial, including 14 days following the last dose of investigational product
* Is currently a user of any illicit drugs (including any marijuana use) or has a history of drug (including alcohol) abuse within approximately 5 years
* has other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or blinded investigational product administration

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 84 clinical trial sites in Australia, Colombia, Guatemala, Israel, Spain, New Zealand, and in the United States. Five hundred participants were screened and 176 randomized.
Groups:
- MK-8521 180 μg: Participants receive double-blind MK-8521 180 μg daily (QD), subcutaneously, over 12 weeks.
- MK-8521 300 μg: Participants receive double-blind MK-8521 300 μg, QD, subcutaneously, over 12 weeks.
- Placebo: Participants receive matching double-blind placebo QD over 12 weeks.
- Liraglutide 1.8 mg: Participants receive open-label liraglutide, 1.8 mg QD, subcutaneously, over 12 weeks.
Period: Overall Study
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Started | 46 | 44 | 43 | 43
Treated | 46 | 44 | 43 | 42
Completed | 30 | 29 | 33 | 30
Not Completed | 16 | 15 | 10 | 13
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0
Not completed — Adverse Event | 3 | 1 | 1 | 2
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Hyperglycemia Discontinuation Criteria | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Non-Compliance With Study Drug | 0 | 1 | 0 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 13 | 10 | 6 | 10

BASELINE CHARACTERISTICS:
Population: All participants randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg | Total
Number analyzed (Participants) | 46 | 44 | 43 | 43 | 176
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (7.6) | 54.2 (7.9) | 51.5 (10.1) | 52.9 (9.4) | 53.2 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 18 | 24 | 20 | 88
  Male | 20 | 26 | 19 | 23 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 2 | 4 | 13
  Asian | 2 | 3 | 4 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 9 | 12 | 7 | 36
  White | 27 | 25 | 23 | 31 | 106
  More than one race | 5 | 4 | 2 | 1 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Hemoglobin A1C Classification by Levels [Number; unit: Participants] — Hemoglobin A1C classification by levels: <8.5% or >=8.5%
  Participants
    <8.5% | 22 | 24 | 24 | 21 | 91
    >=8.5% | 24 | 20 | 19 | 22 | 85
Antihyperglycemic agent (AHA) Washout Status [Number; unit: Participants] — AHA washout status (yes/no). The trial included an 8-week AHA washout period for participants taking a AHA.
  Participants
    Yes | 5 | 5 | 5 | 5 | 20
    No | 41 | 39 | 38 | 38 | 156
Body Mass Index (BMI) [Number; unit: Participants] — Number of participants with a BMI <30 kg/m^2 or BMI>=30 kg/m^2
  Participants
    <30 kg/m^2 | 18 | 14 | 15 | 15 | 62
    >=30 kg/m^2 | 28 | 30 | 28 | 28 | 114
Heart Rate [Mean (Standard Deviation); unit: Beats/minute] — Population: All randomized participants who had a baseline heart rate value.
  Beats/minute
    number analyzed (Participants) | 46 | 44 | 43 | 42 | 175
    (all) | 72.5 (7.7) | 72.2 (9.9) | 73.8 (8.6) | 74.7 (8.9) | 73.3 (8.8)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 171.4 (41.0) | 175.0 (49.5) | 172.0 (39.2) | 187.5 (44.9) | 176.4 (43.9)
Fasting Low Density Lipoprotein (LDL) Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Population: All randomized participants who had a baseline fasting LDL cholesterol value.
  mg/dL
    number analyzed (Participants) | 42 | 41 | 40 | 40 | 163
    (all) | 103.3 (28.1) | 95.6 (33.8) | 100.5 (42.8) | 93.0 (29.5) | 98.2 (33.9)
Fasting High Density Lipoprotein (HDL) Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Population: All randomized participants who had a baseline fasting HDL cholesterol value.
  mg/dL
    number analyzed (Participants) | 42 | 41 | 40 | 40 | 163
    (all) | 47.4 (12.3) | 41.7 (9.5) | 43.1 (12.0) | 46.8 (13.8) | 44.8 (12.1)
Fasting Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Population: All randomized participants who had a baseline fasting triglycerides value.
  mg/dL
    number analyzed (Participants) | 46 | 44 | 43 | 42 | 175
    (all) | 171.5 (104.6) | 167.1 (79.5) | 168.7 (96.1) | 154.0 (89.5) | 165.5 (92.5)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mm Hg] | 125.1 (10.8) | 126.0 (12.0) | 124.6 (14.3) | 126.3 (11.0) | 125.5 (12.0)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mm Hg] | 76.6 (6.3) | 77.9 (7.4) | 77.6 (8.3) | 78.9 (5.7) | 77.7 (7.0)
Hemoglobin A1C [Mean (Standard Deviation); unit: Percent] | 8.54 (0.82) | 8.43 (0.78) | 8.46 (0.83) | 8.72 (1.03) | 8.54 (0.87)
Body Weight [Mean (Standard Deviation); unit: Kilograms] | 85.4 (18.1) | 89.4 (20.0) | 90.2 (19.0) | 92.4 (16.5) | 89.3 (18.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 12
Description: A1C is the percentage of hemoglobin that has glucose bound to it and is a blood marker used to report average blood glucose levels over prolonged periods of time. A1C is reported as a percentage (%). This change from baseline reflects the Week 12 A1C minus the Week 0 A1C.
Time Frame: Baseline and Week 12
Population: All randomized, treated participants with at least one A1C measurement (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 43 | 42
Percent | -0.82 [-1.16 to -0.49] | -1.05 [-1.41 to -0.69] | -0.44 [-0.80 to -0.08] | -1.42 [-1.77 to -1.07]
Statistical Analysis 1: Comparison: MK-8521 180 μg vs Placebo; Test type: Superiority; p = 0.126, Longitudinal data analysis; Terms for treatment, time, A1C (<8.5%, ≥8.5%), BMI (<30 kg/m^2, ≥30 kg/m^2) and AHA washout status (Yes, No), and the interaction of time by treatment; Difference in Least Squares Means = -0.39, 95% CI 2-sided [-0.88 to 0.11]
Statistical Analysis 2: Comparison: MK-8521 180 μg vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.017, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 0.60, 95% CI 2-sided [0.11 to 1.08]
Statistical Analysis 3: Comparison: MK-8521 300 μg vs Placebo; Test type: Superiority; p = 0.018, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.61, 95% CI 2-sided [-1.12 to -0.10]
Statistical Analysis 4: Comparison: MK-8521 300 μg vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.146, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 0.37, 95% CI 2-sided [-0.13 to 0.87]
Statistical Analysis 5: Comparison: Placebo vs Liraglutide 1.8 mg; Test type: Superiority; p < 0.001, Longitudinal data analysis — Terms for treatment, time, A1C (<8.5%, ≥8.5%), BMI (<30 kg/m^2, ≥30 kg/m^2) and AHA washout status (Yes, No), and the interaction of time by treatment; Difference in the Least Squares Means = -0.98, 95% CI 2-sided [-1.49 to -0.48]

2. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to Week 14
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 43 | 42
Participants | 24 | 29 | 25 | 22

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: as for outcome 2
Time Frame: Up to Week 12
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 43 | 42
Participants | 3 | 1 | 2 | 2

4. Primary Outcome: Number of Participants With an AE of Symptomatic Hypoglycemia
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Hypoglycemia episodes are those with glucose values ≤70 mg/dL (3.9 mmol/L). Symptomatic hypoglycemia episodes were episodes with clinical symptoms reported by the investigator as hypoglycemia and classified as adverse events.
Time Frame: Up to Week 14
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 43 | 42
Participants | 0 | 2 | 1 | 1
Statistical Analysis 1: Comparison: MK-8521 180 μg vs Placebo; Test type: Superiority; p = 0.301, Miettinen & Nurminen method; Difference in % vs Placebo = -2.3, 95% CI 2-sided [-12.1 to 5.6]
Statistical Analysis 2: Comparison: MK-8521 300 μg vs Placebo; Test type: Superiority; p = 0.573, Miettinen & Nurminen method; Difference in % vs Placebo = 2.2, 95% CI 2-sided [-8.1 to 13.2]
Statistical Analysis 3: Comparison: MK-8521 180 μg vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.295, Miettinen & Nurminen method; Difference in % vs Liraglutide = -2.4, 95% CI 2-sided [-12.4 to 5.5]
Statistical Analysis 4: Comparison: MK-8521 300 μg vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.587, Miettinen & Nurminen method; Difference in % vs Liraglutide = 2.2, 95% CI 2-sided [-8.4 to 13.2]

5. Primary Outcome: Change From Baseline in Heart Rate at Week 12
Description: This change from baseline reflects the Week 12 heart rate minus the Week 0 heart rate.
Time Frame: Baseline and Week 12
Population: All randomized, treated participants with at least one heart rate measurement (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats/minute
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 43 | 42
Beats/minute | 5.47 [2.99 to 7.96] | 6.28 [3.72 to 8.84] | -1.42 [-3.92 to 1.07] | 1.63 [-0.88 to 4.14]
Statistical Analysis 1: Comparison: MK-8521 180 μg vs Placebo; Test type: Superiority; Difference in the LS Means vs. Placebo = 6.90, 95% CI 2-sided [3.42 to 10.37] — Terms for treatment, time, A1C (<8.5%, ≥8.5%), BMI (<30 kg/m^2, ≥30 kg/m^2) and AHA washout status (Yes, No), and the interaction of time by treatment; Longitudinal data analysis
Statistical Analysis 2: Comparison: MK-8521 180 μg vs Liraglutide 1.8 mg; Test type: Superiority; Difference in LS Means vs. Liraglutide = 3.84, 95% CI 2-sided [0.35 to 7.33] — [estimate comment as in outcome 5, analysis 1]; Longitudinal data analysis
Statistical Analysis 3: Comparison: MK-8521 300 μg vs Placebo; Test type: Superiority; Difference in LS Means vs. Placebo = 7.70, 95% CI 2-sided [4.17 to 11.23] — [estimate comment as in outcome 5, analysis 1]; Longitudinal data analysis
Statistical Analysis 4: Comparison: MK-8521 300 μg vs Liraglutide 1.8 mg; Test type: Superiority; Difference in LS Means vs. Liraglutide = 4.65, 95% CI 2-sided [1.11 to 8.19] — [estimate comment as in outcome 5, analysis 1]; Longitudinal data analysis

6. Secondary Outcome: Change From Baseline in Body Weight at Week 12
Description: This change from baseline reflects the Week 12 body weight minus the Week 0 body weight.
Time Frame: Baseline and Week 12
Population: All randomized, treated participants with at least one body weight measurement (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 43 | 42
Kilograms | -2.0 [-2.9 to -1.1] | -3.0 [-4.0 to -2.1] | -1.3 [-2.2 to -0.3] | -2.9 [-3.8 to -1.9]
Statistical Analysis 1: Comparison: MK-8521 180 μg vs Placebo; Test type: Superiority; p = 0.285, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.7, 95% CI 2-sided [-2.0 to 0.6]
Statistical Analysis 2: Comparison: MK-8521 180 μg vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.183, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 0.9, 95% CI 2-sided [-0.4 to 2.2]
Statistical Analysis 3: Comparison: MK-8521 300 μg vs Placebo; Test type: Superiority; p = 0.010, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.8, 95% CI 2-sided [-3.1 to -0.4]
Statistical Analysis 4: Comparison: MK-8521 300 μg vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.811, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.2, 95% CI 2-sided [-1.5 to 1.2]
Statistical Analysis 5: Comparison: Placebo vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.018, Longitudinal data analysis — [p-value comment as in outcome 1, analysis 5]; Difference in the Least Squares Means = -1.6, 95% CI 2-sided [-2.9 to -0.3]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 12
Description: This change from baseline reflects the Week 12 FPG minus the Week 0 FPG.
Time Frame: Baseline and Week 12
Population: All randomized, treated participants with at least one FPG measurement (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 43 | 42
mg/dL | -13.7 [-27.7 to 0.3] | -34.6 [-49.3 to -19.9] | -5.1 [-19.4 to 9.2] | -42.9 [-57.0 to -28.7]
Statistical Analysis 1: Comparison: MK-8521 180 μg vs Placebo; Test type: Superiority; p = 0.385, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -8.6, 95% CI 2-sided [-28.2 to 10.9]
Statistical Analysis 2: Comparison: MK-8521 180 μg vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.004, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 29.1, 95% CI 2-sided [9.7 to 48.6]
Statistical Analysis 3: Comparison: MK-8521 300 μg vs Placebo; Test type: Superiority; p = 0.004, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -29.5, 95% CI 2-sided [-49.6 to -9.4]
Statistical Analysis 4: Comparison: MK-8521 300 μg vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.416, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 8.3, 95% CI 2-sided [-11.7 to 28.2]
Statistical Analysis 5: Comparison: Placebo vs Liraglutide 1.8 mg; Test type: Superiority; p < 0.001, Longitudinal data analysis — [p-value comment as in outcome 1, analysis 5]; Difference in the Least Squares Means = -37.8, 95% CI 2-sided [-57.5 to -18.0]

8. Secondary Outcome: Change From Baseline in Fasting Low Density Lipoprotein (LDL) Cholesterol at Week 12
Description: This change from baseline reflects the Week 12 fasting LDL cholesterol minus the Week 0 fasting LDL cholesterol.
Time Frame: Baseline and Week 12
Population: All randomized, treated participants with at least one fasting LDL cholesterol measurement (baseline or post-baseline).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Number analyzed (Participants) | 27 | 26 | 28 | 29
mg/dL | -9.3 (23.5) | 8.8 (41.8) | 4.5 (33.5) | 0.3 (18.0)

9. Secondary Outcome: Change From Baseline in Fasting High Density Lipoprotein (HDL) Cholesterol at Week 12
Description: This change from baseline reflects the Week 12 fasting HDL cholesterol minus the Week 0 fasting HDL cholesterol.
Time Frame: Baseline and Week 12
Population: All randomized, treated participants with at least one fasting HDL cholesterol measurement (baseline or post-baseline).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Number analyzed (Participants) | 27 | 26 | 28 | 29
mg/dL | -0.4 (12.3) | -0.5 (6.0) | 3.8 (6.6) | 0.4 (5.7)

10. Secondary Outcome: Change From Baseline in Fasting Triglycerides at Week 12
Description: This change from baseline reflects the Week 12 fasting triglycerides minus the Week 0 fasting triglycerides.
Time Frame: Baseline and Week 12
Population: All randomized, treated participants with at least one fasting triglycerides measurement (baseline or post-baseline).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Number analyzed (Participants) | 31 | 27 | 31 | 30
mg/dL | -2.9 (91.9) | -26.6 (71.2) | -15.6 (68.9) | -20.5 (48.6)

11. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Week 12
Description: This change from baseline reflects the Week 12 SBP minus the Week 0 SBP.
Time Frame: Baseline and Week 12
Population: All randomized, treated participants with at least one SBP measurement (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 43 | 42
mmHg | -2.7 [-6.4 to 0.9] | -1.5 [-5.2 to 2.3] | 1.0 [-2.6 to 4.6] | -1.7 [-5.3 to 2.0]
Statistical Analysis 1: Comparison: MK-8521 180 μg vs Placebo; Test type: Superiority; p = 0.151, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -3.7, 95% CI 2-sided [-8.8 to 1.4]
Statistical Analysis 2: Comparison: MK-8521 180 μg vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.682, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.1, 95% CI 2-sided [-6.2 to 4.1]
Statistical Analysis 3: Comparison: MK-8521 300 μg vs Placebo; Test type: Superiority; p = 0.344, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -2.5, 95% CI 2-sided [-7.7 to 2.7]
Statistical Analysis 4: Comparison: MK-8521 300 μg vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.948, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 0.2, 95% CI 2-sided [-5.0 to 5.4]
Statistical Analysis 5: Comparison: Placebo vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.306, Longitudinal data analysis — [p-value comment as in outcome 1, analysis 5]; Difference in the Least Squares Means = -2.7, 95% CI 2-sided [-7.8 to 2.5]

12. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at Week 12
Description: This change from baseline reflects the Week 12 DBP minus the Week 0 DBP.
Time Frame: Baseline and Week 12
Population: All randomized, treated participants with at least one DBP measurement (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 43 | 42
mmHg | 0.5 [-1.7 to 2.8] | 0.4 [-1.9 to 2.8] | -1.0 [-3.3 to 1.3] | 0.6 [-1.7 to 2.9]
Statistical Analysis 1: Comparison: MK-8521 180 μg vs Placebo; Test type: Superiority; p = 0.347, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 1.5, 95% CI 2-sided [-1.7 to 4.8]
Statistical Analysis 2: Comparison: MK-8521 180 μg vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.963, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.1, 95% CI 2-sided [-3.3 to 3.2]
Statistical Analysis 3: Comparison: MK-8521 300 μg vs Placebo; Test type: Superiority; p = 0.394, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 1.4, 95% CI 2-sided [-1.9 to 4.7]
Statistical Analysis 4: Comparison: MK-8521 300 μg vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.905, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.2, 95% CI 2-sided [-3.5 to 3.1]
Statistical Analysis 5: Comparison: Placebo vs Liraglutide 1.8 mg; Test type: Superiority; p = 0.325, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in the Least Squares Means = 1.6, 95% CI 2-sided [-1.6 to 4.9]

ADVERSE EVENTS:
Time Frame: Up to Week 14
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The analysis population included all treated participants.
Arm/Group | MK-8521 180 μg | MK-8521 300 μg | Placebo | Liraglutide 1.8 mg
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/44 | 1/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/46 | 1/44 | 1/43 | 0/42
Other Adverse Events (participants affected / at risk) | 18/46 | 21/44 | 15/43 | 13/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8521 180 μg (N=46) | MK-8521 300 μg (N=44) | Placebo (N=43) | Liraglutide 1.8 mg (N=42)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8521 180 μg (N=46) | MK-8521 300 μg (N=44) | Placebo (N=43) | Liraglutide 1.8 mg (N=42)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 3 (3) | 1 (2) | 3 (4)
Nausea (Gastrointestinal disorders) | 6 (8) | 7 (10) | 1 (1) | 9 (12)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 1 (1) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 3 (5) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 3 (5) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 4 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT02492763/Prot_SAP_000.pdf